CLINICAL TRIAL: NCT05505266
Title: Physical Activity, Quality of Life, Emotional State and Coping Strategies in Climacteric Women.
Brief Title: Physical and Emotional Coping Variables in Climacteric Women
Acronym: ClimWo
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Other Study IDs: ID0037
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Menopausal Women
Keywords: climateric women
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — observational

SUMMARY:
Introduction: The transition to menopause entails several changes in the biopsychosocial sphere of climacteric women. Compared to other therapies, physical exercise has no side effects, is not costly and can have a positive influence on the symptoms reported by women at this stage. The emotional and physical state of climacteric women is affected by the alterations typical of menopause, deteriorating their quality of life. Likewise, physical exercise improves the associated symptomatology. The objective is to know how the study variables (symptomatology, quality of life, emotional state, physical exercise and level of coping) correlate.

Material and methods: Cross-sectional descriptive observational design with a study population made up of women in the climacteric stage carried out through an anonymous and voluntary survey.

DETAILED DESCRIPTION:
The climacteric is a progressive period, which lasts for years, before and after menopause, the latter being the physiological stage of aging characterized by the decrease in the follicular function of the ovaries that ends with the cessation of menstrual periods. permanent, a phenomenon associated with the decrease in the production of hormones, as well as the arrest by the ovaries in the release of ovules. Menopause most commonly occurs between the ages of 45 and 55. The climacteric is experienced by each woman in a different way, since it is also influenced by biopsychosocial factors, but the investigators can speak of a common symptomatology typical of the climacteric that groups together vasomotor symptoms such as hot flashes and palpitations, psychological symptoms such as changes in mood, depression, irritability and anxiety, alterations in sleep quality, cognitive symptoms such as memory loss, among others. Among the therapies to alleviate the symptoms associated with menopause, the investigators find estrogenic and non-estrogenic hormonal therapies, inhibitors and physical exercise.

Despite the lack of evidence to support physical exercise as a tool to eradicate symptoms linked to menopause, the investigators can affirm that it relieves both somatic and psychological symptoms, and vasomotor and sexual symptoms to a lesser extent, which is associated with an improvement overall quality of life. In addition, with regular physical activity the investigators will be able to strengthen the musculoskeletal system and improve the quality of life.

The investigators found a scarcity of studies that relate therapeutic exercise as a physiotherapeutic tool in relieving the symptomatology of climacteric women, for this reason the need to study the activity they carry out in this area and know its characteristics is raised, in order to guide future strategies in physiotherapy.

Objective: To know the physical exercise carried out by women in this period, to know the existence of levels of anxiety and depression, Coping level and quality of life.

Material and methods Subjects: Women between 40 and 60 years old. For the development of the study, a questionnaire is prepared, which consists of an initial section with basic questions about personal data and symptomatology referred to by each subject, to later move on to the rest of the sections that will include questions from other validated questionnaires: quality of life using the SF -12; For the emotional state, the Goldberg scale; For physical activity, the International Physical Activity Questionnaire (IPAQ); And for coping level, the Brief COPE inventory.

At the end, 2 questions are included about how often they go to a physical therapist to deal with musculoskeletal pain.

Once the questionnaire is closed, the results will be analyzed using SPSS, which will allow us to contrast hypotheses and generate new ones.

ELIGIBILITY:
Inclusion Criteria:

* Climacteric women
* Age between 40 and 60 years.

Exclusion criteria:

- Not having internet access to complete the questionnaire.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — climacteric women
Study Population: Climacteric women
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Physical activity | 1 day
  It is evaluated using the International Physical Activity Questionnaire (IPAQ). This questionnaire in its short version consists of 7 questions about the frequency, duration and intensity of physical activity performed during the last 7 days and is designed to be used with adults between the ages of 18 and 65. The aim is thus to monitor the time spent for each type of activity. Weekly physical activity will be quantified in Metabolic Rate Units (METs) per minute and per week. The reference values used in this questionnaire mark 3.3 METs for walking, 4 METs for moderate physical activity and 8 METs for intense physical activity. These amounts must be multiplied by the time in minutes and by the number of days used to carry out each of the different exercise modalities according to their value. The IPAQ classifies the level of physical activity performed into 3 categories: low, medium and high.

SECONDARY OUTCOMES:
Well-being | 1 day
  It is evaluated using the SF-12 questionnaire. This questionnaire thus provides an instrument to assess the functional capacity and level of well-being of people over 14 years of age, in order to define a positive or negative state of physical and mental health, testing for each of them 4 dimensions, resulting in a total of 8 different dimensions in the entire questionnaire, which are mentioned below: for physical health; physical function, physical role, bodily pain and general health and for mental health; social function, emotional role, mental health and vitality. The response modality for each of the questions is Likert-type, that is, the scales have between 3 and 6 points, depending on the number of options. They aim to assess the intensity and/or frequency of the degree of health of the women surveyed. The total score of the questionnaire is collected between the values 0 and 100, being a high score equivalent to a better health condition of the person.
Anxiety and depression | 1 day
  It is evaluated using the Goldberg Anxiety and Depression Scale (GADS). In the test, questions are asked that refer to the state of mind of the last 2 weeks, with questions about the symptoms mentioned, specifically, 4 will be specific to anxiety and another 4 specific to depression. Given 2 or more affirmative answers in the anxiety section, another 5 questions about anxiety will be asked and, following the same line, if 1 or more positive answers are obtained in the depression section, the test will end with 5 more questions.This means that, if at least 2 affirmative questions were obtained from the 4 existing anxiety questions and 1 affirmative question from depression questions, we would have that the scale consists of a total of 18 questions, with 9 in each subscale. The cut-off points assigned to classify the existence of anxiety are 4 or more points, which are obtained with each affirmative answer, and 2 or more points to classify depression.
Coping level | 1 day
  It is evaluated through the COPE-28 inventory. This inventory consists of 28 questions, with 2 items for each of the 14 subscales. It has four response alternatives, scored from 0 to 3, which refer to "I never resort to this" to "I always resort to this" with intermediate scores; "almost never" and "frequently". Once the inventory is complete, the score of two items of each subscale will be added. High scores indicate more frequent use of that coping style.
  This questionnaire collects the following variables: active coping, emotional support, social support, self-blame, acceptance, self-distraction, relief, behavioral disconnection, humor, denial, planning, positive reinterpretation, religion, and use of substances such as alcohol or medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma V Espí-López, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No